CLINICAL TRIAL: NCT05544955
Title: Comparison of Protein Ingestion Timing on Body Composition, Physical Performance, and Biochemical Markers in Resistance-trained Males
Brief Title: Protein Ingestion Timing on Body Composition and Biochemical Markers in Resistance-trained Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marymount University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexei Wong, Associate Professor, Marymount University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IR.SSRC.REC.1403.059
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophy; Physical Performance
MeSH Terms: conditions — Hypertrophy | interventions — Lead

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein ingestion immediately prior to and immediately after resistance training (Experimental): This arm involved protein ingestion immediately prior to and immediately after resistance training for 12 weeks. Participants will consume 40 g of isolate whey protein at their recommended timing.
  Interventions: Dietary Supplement: isolate whey protein prior to and immediately after resistance training
- Protein ingestion 3 hours prior to and 3 hours after resistance training (Experimental): This arm involved protein ingestion 3 hours prior to and 3 hours after resistance training for 12 weeks. Participants will consume 40 g of isolate whey protein at their recommended timing.
  Interventions: Dietary Supplement: isolate whey protein 3 hours prior to and 3 hours after resistance training

INTERVENTIONS:
Dietary Supplement: isolate whey protein prior to and immediately after resistance training — This arm involved protein ingestion immediately prior to and immediately after resistance training for 12 weeks. Participants will consume 40 g of isolate whey protein at their recommended timing.
  Arms: Protein ingestion immediately prior to and immediately after resistance training
Dietary Supplement: isolate whey protein 3 hours prior to and 3 hours after resistance training — This arm involved protein ingestion 3 hours prior to and 3 hours after resistance training for 12 weeks. Participants will consume 40 g of isolate whey protein at their recommended timing.
  Arms: Protein ingestion 3 hours prior to and 3 hours after resistance training

SUMMARY:
Protein ingestion timing is an important component for muscle accretion. The investigators hypothesized that protein ingestion timing could affect muscular adaptations and performance in resistance-trained men.

ELIGIBILITY:
Inclusion Criteria:

* performing resistance training at least three times a week for 1 year prior to the start of the study
* not taking any steroids or any illegal agents known to increase muscle size for at least 1 year prior to the start of the study
* no known medical issues
* sleeping for at least seven to eight hours during the 24-hour day

Exclusion Criteria:

* non-willingness to continue protein ingestion or exercise protocols
* participation in exercise other than the prescribed resistance training program
* consumption of dietary supplement (other than the protein intervention) during the study period
* Missing more than one resistance training session or protein ingestion throughout the study period

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Body Composition | 12 weeks
  Total Lean mass, fat mass, and estimated VAT (g) will be assessed using whole-body DXA

SECONDARY OUTCOMES:
Muscular Strength | 12 weeks
  Using 1 repetition maximum
Muscular Endurance | 12 weeks
  Using leg- and chest press exercises at 75% of the 1-RM
Jump testing | 12 weeks
  Using the vertical and broad jump tests
Pull-ups | 12 weeks
  Using the pull-up test
Liver enzymes (ALT, AST, and GGT) | 12 weeks
  Using Fasting blood samples
Creatinine and Urea Nitrogen | 12 weeks
  Urine samples will be collected using standard procedures
Cholesterol Levels | 12 weeks
  Using Fasting blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Marymount University, Arlington, Virginia, United States